CLINICAL TRIAL: NCT01232673
Title: Autologous Bone Marrow Stem Cell Transfer in Patients With Chronical Critical Limb Ischemia and Diabetic Foot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-99/OVZ/08/006-Dot
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia; Bone-Marrow Aspiration Concentrate; Diabetes Mellitus; Major Amputation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetes Mellitus | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMAC treatment active group (Experimental): Collection of 240ml from both illiac crests, followed by gradient density centrifugation, resulting in obtaining 40ml of BMAC. This ammount is applied by one ml per injection into the critical limb ischemia along the calf vessels.
  Interventions: Procedure: BMAC application in Critical Limb Ischemia
- Control Study Group (No Intervention): Standard treatment group of patients with CLI after surgical or interventional revascularisation will serve as control.

INTERVENTIONS:
Procedure: BMAC application in Critical Limb Ischemia — Collection of 240ml from both illiac crests, followed by gradient density centrifugation, resulting in obtaining 40ml of BMAC (Bone-Marrow Aspiration Concentrate). BMAC is subsequently administered into the ischemic limb along calf vessels.
  Other Names: Critical Limb Ischemia; Bone-Marrow Aspiration Concentrate; Laser Doppler
  Arms: BMAC treatment active group

SUMMARY:
A total of 90 patients suffering from end stage-IV Fontaine /CLI and diabetic foot with an ulcerated limb in whom all previous therapeutic strategies failed (e.g. surgical revascularization) will be selected and undergo local transplantation of ABMSCs. The efficacy/safety of this therapy will be assessed by using several endpoints such as (a) prevention of amputation, (b) wound healing and (c) degree of angiogenesis. In order to assess the limb ischemia and hypoxia the several tests and measurements will be performed pre- and post transplantation at a variety of time intervals. The measurements include: TP-toe pressure measurements (by Periflux 5000 Laser Doppler and Oxymetry system), SPP-skin perfusion pressure, ABI-ankle brachial index, LDP-laser Doppler baseline and heat perfusion assessment, TcpO2 without and with O2 provocation inhalation test. In addition, a battery of biochemical and hematological tests of peripheral venous blood sample will be performed.The quality form "EQ-50" will be completed.

8.1 Primary objective: To evaluate an efficacy-safety profile of autologous bone marrow stem cells (ABMSCs) transplantated into chronically and critically ischemic limb (CLI) and into diabetic foot in stage IV Fontaine, Rutherfod 4-6 classification.

8.2 Secondary objectives: 8.2.1 To assess effect of ABMSCs on tissue perfusion of ischemic limb after transplantation by transcutaneous oximetry and the laser Doppler flowmetry using Periflux 5000 system under normal and provocation test conditions. In addition, wound healing of ulcers will be evaluated using a planimetry method from photographs of affected skin taken pre- and post-transplantation.

8.2.2 Relationship between CD 34 progenitor counts separated on gradient-density separation centrifuge from Harvest Technologies and overall effectiveness and safety to treat ischemic limb.

8.3 Priorities: Beside assessment of effectiveness and safety of ABMSCs transplantation ultimate emphasis will be put on avoiding limb amputation. This has significant socioeconomic impact. Therefore this project belongs to the priority programs of clinical research in cardiovascular diseases.

DETAILED DESCRIPTION:
1. INTRODUCTION:

   The local method of autologous bone marrow stem cells transplantation consists of harvesting bone marrow from the iliac crest, its separation using cell separator to generate ABMSCs (CD 34 positive) and their subsequent multiple injections into a limb suffering from chronic and critical ischemia. The aim of this therapy is to induce angiogenesis and vasculogenesis which would correct ischemia and hypoxia, improve tissue perfusion and metabolism and thus prevent limb amputation. Due to correction of hypoxia and ischemia by improvement of blood supply regeneration of damaged tissues is initiated. Improved tissue perfusion is achieved by a large number of mediators including growth and angiogenic factors which in turn stimulate growth of primitive vessel wall within the ischemic tissue, a part of healing process. In general, such reparative process could be divided into the initial phase characterized by the release of inflammatory mediators and neurotransmitters followed by phase of formation of primitive vascular tubes composed of the endothelial cell precursors which are later on adhered to and stabilized by pericyte cells. Process of angiogenesis (by sprouting as well as nonsprouting) takes usually between 4-6 weeks depending on degree of the initial tissue ischemia and hypoxia. Development of new collateral blood flow in the ischemic/hypoxic tissue can be monitored by the Laser Doppler - Flowmetry, level of Transcutaneous TcpO2 and TcpCO2, Toe Pressure and Skin Perfusion Pressure measurements, the Index Ankle-Arm ABI using Duplex Doppler Ultrasound, angiography, MRI or alternatively by common methods used in nuclear medicine. Analysis and interpretation of all these measurements should define degree of efficacy and safety of this therapeutic modality and may suggest future directions in optimization of this therapy.
2. PROJECT OBJECTIVES:

Primary objective: To evaluate an efficacy-safety profile of autologous bone marrow stem cells (ABMSCs) transplantated into chronically and critically ischemic limb (CLI) and into diabetic foot in stage IV Fontaine classification.

Secondary objectives: To assess effect of ABMSCs on tissue perfusion of ischemic limb after transplantation by transcutaneous oximetry and the laser Doppler flowmetry using Periflux 5000 system under normal and provocation test conditions. In addition, wound healing of ulcers will be evaluated using a planimetry method from photographs of affected skin taken pre- and post-transplantation.

Relationship between CD 34 progenitor counts separated on gradient-density separation centrifuge from Harvest Technologies and overall effectiveness and safety to treat ischemic limb.

Priorities: Beside assessment of effectiveness and safety of ABMSCs transplantation ultimate emphasis will be put on avoiding limb amputation. This has significant socioeconomic impact. Therefore this project belongs to the priority programs of clinical research in cardiovascular diseases.

METHODOLOGY AND PATIENT RECRUITMENT:

A total of 90 patients (45 patients per year) will be recruited over the period of 2 years for this study.

Separation of ABMSCs and their application:

Concentrate of autologous stem cells (CD 34 positive) will be separated from the bone marrow aspirate using the cell separator from Harvest Technologies. Bone marrow is collected from both iliac bone shovels according to standard Yamshidi puncture aspiration methodology. During this procedure the patient is under analgosedation using propophol iv bolus and physiological signs including blood pressure (BP), pulse, ECG, pO2 saturation are continuously monitored and adjusted according to needs. In brief, 240 ml of the bone marrow is aspirated into an aspiration set pre filed with ACD-A anticoagulant (30 ml) by hematologist and processed using the cell separator from Harvest Technologies. This equipment is easy to operate and has several advantages compared to other cell separators on the market. The methodology is (a) simple, easy, fast, and safe using gradient density centrifugation to separate all blood elements including white cells, platelets, red cells from collected bone marrow in centrifuge containers into a sample with 5 % hematocrit (containing ABMSCs and platelets) within 15 minutes. Thereafter 40 ml of sample is aspirated into a syringe and immediately applied by multiple injections in the ischemic limb. Whole procedure should take less than one hour.

Monitoring of quality and clinical effects of ABMSCs transplantation:

Bone marrow will be examined before and after separation of ABMSCs to assess number of CD 34 positive progenitors as well as number of other cellular components including platelets. Prior- (0 days-baseline) and post transplantation (1, 7, 14, 30, 60, and 120 days) all patients will undergo following examinations: Laser Doppler Flowmetry - assessment of blood flow; measurements of transcutaneous oxygen (TcpO2) and CO2 (TcpCO2) levels with and without provocation test (with O2 inhalation). Complete battery of tests such as CBC and differential, fibrinogen and CPR will also be established. In addition, ABI-Ankle-Brachial Index, TP-Toe Pressure, SPP-Skin Perfusion Pressure, Rutherford and Fontaine Cathegory, analgetics consumption (requirements), claudication interval in non-amputated patients will also be monitored. These values will be collected and then correlated with the degree of initial ischemia/hypoxia as well as with changes in ischemia/hypoxia developed within 120 postoperative days (6 intervals).

4 / EXPECTED RESULTS AND THE IMPORTANCE OF SOCIO-ECONOMIC IMPACT Our preliminary pilot data suggest that in 60% of patients suffering from chronic critical limb ischemia which failed to common therapy, limb amputations were prevented. In this patients leg wound healed very well within the 120 days following ABMSCs transplantation. This is a remarkable success when compared to historical controls with 100% amputations, particularly in ischemic leg at the end-stages with failed therapy (Rutherford 4-6 and Fontaine IV classification) of CLI and diabetic foot with wounds. We expect to confirm these results and set a new standard for the treatment of this condition with ABMSCs transplantation in Faculty Hospital Ostrava and the Czech Republic as well. We feel that our new treatment will have significant positive socioeconomic impact on our patients and entire Czech society.

5 / MATERIALS AND HUMAN RESOURCES 5.1 Patients included in the project will be examined in the interventional angiology FN Ostrava laboratory were inclusion end exclusion criteria will be considered. They will be included to the study after completing standard revascularisation (Bypass or PTA-stent of the leg arteries) treatment, meeting the criteria of end-stage Fontaine - IV and Rutherford 4-6 classification of the CLI.

5.2 Entrance examinations - will be carried out by the duplex doppler legs examination, measuring of ankle pressure, ankle-brachial index and toe pressure, measurement of SPP- skin perfusion pressure with laser doppler and measurement of transcutaneous TcpO2 and TcpCO2. The patient will have initial angiographic examination by DSA, CTA or MRA to assess depleted basic revascularisation treatment.

5.3 Personnel cooperation: The candidate -Vaclav Prochazka, MD, PhD, MSc will coordinate patients recruitment, entry examinations carry out and will be involved in data collection and data management. Jaromir Gumulec, MD will participate in the bone marrow collection and separation and data-processing, blood samples laboratory tests and data management. Prof.. Peter Klement, MVDr, Ph.D. will contribute to ensure the logistics and processing of statistical datas and ensure the publications and presentations in the foreign journals. Frantisek Jaluvka, MD will contribute patients hospitalisation to the surgical clinic, subsequent podology ambulatory care for these patients and will participate in the BMSC transplantatation procedure to ensure desinfection and sterility of operating environment. Jana Chmelova, MD. will participate on the transplantation programe procedures, data processing and ensuring the creation of publications.

6 / TIME WORK PLAN During the first and second year 45 patients each will be enrolled (in total 90). All patients will be treated with autologous BMSC Tx and monitoring of clinical state with endpoints of limb amputation or wound healing will be donne. Hematology datas of separated bone marrow samples will be analysed and examination of peripheral venous blood samples laboratory datas at day 0,1,3,7,14,30 will be carried out. Entire datas of tissue perfusion with laser doppler flow (LDP), including provocation tests and measurements of TcpO2 and TcpCO2 including inhalation tests for appreciation of the tissue perfusion state will be evaluated. Ankle pressures with the ABI- index, SPP- skin perfusion pressure and TP- toe pressure will be examined. Simultaneously dynamic legs scintigraphy before and 6 months after the procedure will be carried out. In the non-amputated patients claudication interval will be tested and Rutherford plus Fontaine stage classification will be counted. In the last 3rd year of the project, patients follow-up will continue with data files and statistical evaluation managements. In the 1st. and 2nd year, interim period report with the economic data assessment will be taken out and in the 3rd year final report will be completed.

7 / INFORMED CONSENT Dear patient Mr/Mrs.., You have been invited by Your doctor for the therapeutic procedure of autologous bone marrow stem cells transplantation. You have the right to freely decide on about further proposed procedure (if specific legislation do not exclude this right) and you have the inalienable right to be fully informed about these procedure. Based on Your current health status, therapeutic procedure of the bone marrow stem cells transplantation for the treatment of chronical critical limb ischemia was designed to You by Your medical specialist.

8 / CONCLUSION OF THE PROJECT The project will be prepared for publication in the Circulation and Stem Cell Therapy journals and will be presented at domestic and foreign angiology, haematology and vascular surgery meetings, with the publication of abstracts accompanied by IGA grant annotations.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from chronic and critical limb ischemia according to the TASC classification Rutherford 4-6, Fontaine IV,
* with failed basic conservative and revascularization treatment (surgical or endovascular),
* with age over 18 years,
* with signed informed consent for this procedure,
* without acute CLI that would require early limb amputation.

Exclusion Criteria:

* patients with estimated survival less than 6 months,
* with known bone marrow diseases,
* with the final stage of renal failure and dialysed,
* with acute stage of severe limb ischemia with severe inflammatory process affecting patient's life which require limb amputation to avert deterioration in clinical condition and death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Major limb amputation | 120 days
  The measure is the number of major limb amputations within 120 days from the procedure.

SECONDARY OUTCOMES:
Tissue perfusion measurements | 120 days
  Measurements of circulatory and blood parameters by laser Doppler flowmetry (TCPO2, TCPCO2, ankle-brachial index - ABI, toe-pressure-TP, toe-brachial index-TBI, skin-persusion pressure-SPP. Peripheral blood tests - white blood cell counts, differention counts, fibrinogen CRP and platelet counts. Bone marrow concentrate analysis to assess the number of CD34 progenitor cells, PQ-50 quality of life questionnaire. Follow-up angiogrwaphy at 120 postoperative days, wound healing measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Vaclav Prochazka, MD, PhD, Principal Investigator — University Hospital Ostrava

REFERENCES:
- [Result] Prochazka V, Gumulec J, Jaluvka F, Salounova D, Jonszta T, Czerny D, Krajca J, Urbanec R, Klement P, Martinek J, Klement GL. Cell therapy, a new standard in management of chronic critical limb ischemia and foot ulcer. Cell Transplant. 2010;19(11):1413-24. doi: 10.3727/096368910X514170. Epub 2010 Jun 7. PMID 20529449